CLINICAL TRIAL: NCT07169786
Title: The Association Between Dietary Pattern and the Progression of Chronic Kidney Disease in Patients With Type 2 Diabetes Mellitus
Brief Title: Diet and Progression of CKD in Patients With Type 2 Diabetes Mellitus
Status: Not yet recruiting | Type: Observational
Sponsor: Mariam Emeel Haleem Naseem (Other)
Responsible Party: Sponsor-Investigator, Mariam Emeel Haleem Naseem, resident physician ,internal medicine, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Diet effect on CKD Type 2 DM
Record Dates: First submitted 2025-08-22; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: CKD Stage 1-4; Diet Pattern Analysis; Type2 Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the relationship between dietary patterns and the progression of chronic kidney disease (CKD) in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a prevalent and serious complication among patients with type 2 diabetes mellitus (T2DM), affecting up to 40% of diabetic individuals and significantly contributing to morbidity and mortality . The interplay between T2DM and CKD is complex, with diabetic kidney disease (DKD) representing a leading cause of end-stage renal disease worldwide Diet is a modifiable risk factor with a profound impact on both the development and progression of CKD in patients with T2DM. Western dietary patterns, characterized by high intakes of salt, saturated fat, red and processed meats, and refined sugars, are associated with increased risk of hypertension, glomerular damage, and accelerated kidney dysfunction.

Conversely, diets rich in vegetables, fruits, whole grains, fiber, legumes, and plant-based proteins have been linked to protective effects against CKD progression. For instance, moderate vegetable protein intake appears to offer renal protection, while excessive consumption of red and processed meats burdens the kidneys and accelerates dysfunction Dietary recommendations should be individualized, taking into account disease severity, comorbidities, and patient preferences This study will investigate the relationship between dietary patterns and the progression of chronic kidney disease (CKD) in patients with type 2 diabetes mellitus The aim of this study is to investigate the relationship between dietary patterns and the progression of chronic kidney disease (CKD) in patients with type 2 diabetes mellitus. This study seeks to

1. Assess how different types of diets (e.g., Mediterranean, DASH, plant-based, high-protein, low-protein) influence the rate of CKD progression in individuals with T2DM.
2. Evaluate the impact of specific dietary components-such as protein and sodium intake-on renal function markers, including estimated glomerular filtration rate (eGFR) and albuminuria, in this patient population.
3. Identify dietary factors that may be protective or detrimental to kidney health in patients with T2DM, with the goal of informing evidence-based dietary recommendations for slowing CKD progression Methodology 2.4.1- Type of the study cross-sectional, observational study

   2.4. 2- Study Setting: The study will be conducted in the internal medicine department in Assiut University hospital.

   2.4. 3- Study subjects:
   1. Inclusion criteria:

      • Adults aged above 18 years
      * Diagnosed with type 2 diabetes mellitus according to ADA criteria.
      * Diagnosed with chronic kidney disease stages 1-4 (eGFR 15-90 mL/min/1.73 m²) for at least 3 months.
      * Willing and able to provide informed consent.
   2. Exclusion criteria:

      • Patients with end-stage renal disease (CKD stage 5 or on dialysis).

      • History of kidney transplantation.

      • Acute kidney injury within the past 3 months.

      • Pregnant or lactating women.
      * Patients with severe comorbid conditions (e.g., active malignancy, severe heart failure).
      * Use of medications known to significantly affect renal function (other than standard antihypertensive or antidiabetic therapy).
   3. Sample Size Calculation:

      Based on determining the main outcome variable, The estimated minimum required sample size is 160 patients .

      The sample size was calculated using Epi-info version 7 software, based on the following assumptions:

      Main outcome variable is to investigate the relationship between dietary patterns and the progression of chronic kidney disease (CKD) in patients with type 2 diabetes mellitus. Based on previous studies [5], Approximately 30% to 40% of patients with T2DM are estimated to have CKD, and based on the percentage confidence limits of 5% and a Confidence level=90% .

      2.4.4 -Study tools:

      Data Collection:

      • Medical History and Demographics: Collection of demographic data (age, sex, ethnicity, education, socioeconomic status), detailed medical history (duration of diabetes, comorbidities such as hypertension and cardiovascular disease, family history, and medication use).

      • Physical Examination: Standardized measurement of height, weight, body mass index (BMI), waist circumference, and blood pressure. Blood pressure will be measured using a calibrated automated sphygmomanometer, with the average of two readings taken after five minutes of rest.

      • Dietary Assessment:

      To comprehensively evaluate dietary intake and patterns:

      • Food Frequency Questionnaire (FFQ): Participants will complete a validated FFQ specifically adapted for the local population and suitable for all age groups. The FFQ will capture habitual dietary intake and will include a broad range of food groups such as refined grains, whole grains, legumes, cruciferous and leafy vegetables, tubers, fungi, fruits, red and processed meats, poultry, fish and seafood, dairy products, eggs, snacks, and fast foods.

      Frequency of consumption will be recorded using standardized categories (never/rarely, 1-2 days/week, 3-4 days/week, 5-6 days/week, daily), which will be converted to numerical values for quantitative analysis. The FFQ will be designed to capture both the diversity and frequency of food intake, as well as preparation methods (e.g., frying, steaming, grilling) and portion sizes, using visual aids and standardized household measures to improve accuracy.

      • 24-Hour Dietary Recalls: To enhance the precision of dietary assessment, three non-consecutive 24-hour dietary recalls (including one weekend day) will be conducted to recall of all foods and beverages consumed, including condiments, snacks, and supplements. Portion sizes will be estimated using food models, and standardized measurement tools.

      • Dietary Data Analysis:. Dietary data will be analyzed for macronutrient and micronutrient intake, focusing on protein, sodium, potassium, phosphorus, fiber, and types of dietary patterns (e.g., Mediterranean, DASH, plant-based, etc.).

      Laboratory Methods • Blood Sampling: Fasting blood samples will be collected to measure serum creatinine, urea, albumin, lipid profile (total cholesterol, LDL, HDL, triglycerides), HbA1c, and electrolytes (sodium, potassium, calcium, phosphorus).

      • Urine Sampling: Spot urine samples will be obtained at the same intervals for albumin-to-creatinine ratio (ACR) and proteinuria assessment, following ADA guidelines for CKD monitoring.

      • Renal Function Calculation: Estimated glomerular filtration rate (eGFR) will be calculated using the CKD-EPI formula to monitor kidney function over time.

      Anthropometric and Clinical Measurements • Body Composition: Height, weight, BMI, and waist and mid arm circumference will be measured at each visit using standardized protocols to track changes in body composition and assess obesity-related risk factors.

      • Blood Pressure: Blood pressure will be measured at each visit, to monitor hypertension as a key risk factor for CKD progression and cardiovascular disease.

      Cardiovascular Disease Risk Assessment

      • Medical and Family History: Detailed history of cardiovascular events (myocardial infarction, stroke, angina, heart failure), family history of CVD, and current use of cardiovascular medications will be collected.

      • Electrocardiogram (ECG): Annual ECGs will be performed to detect arrhythmias, ischemic changes, or evidence of prior myocardial infarction, especially in older participants or those with known risk factors.

      • Lifestyle Assessment: Smoking status, alcohol consumption, and physical activity will be recorded. Follow up previous data will be recorded after 6 months

      2.4.5 - Research Outcome Measures • Primary Outcomes Measures • Evaluation of the influence of dietary pattern on the progression of chronic kidney disease among patients with type 2 diabetes mellitus • Prevalence of chronic kidney disease (CKD) among patients with type 2 diabetes mellitus (T2DM), as defined by estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m² and/or albumin-to-creatinine ratio (ACR) ≥30 mg/g at the time of assessment

      • Distribution of CKD stages among T2DM patients at the time of data collection.
      * Secondary outcomes Measures
      * Prevalence of albuminuria and reduced eGFR in the study population
      * Identification and analysis of sociodemographic, clinical, and lifestyle factors associated with the presence of CKD, such as age, sex, duration of diabetes, blood pressure, glycemic control (HbA1c), body mass index (BMI), dietary patterns, and comorbidities (e.g., hypertension, dyslipidemia, cardiovascular disease)
      * Prevalence of cardiovascular risk factors (e.g., hypertension, dyslipidemia, obesity) among T2DM patients with and without CKD

ELIGIBILITY:
Inclusion Criteria:

* • Adults aged above 18 years

  * Diagnosed with type 2 diabetes mellitus according to ADA criteria.
  * Diagnosed with chronic kidney disease stages 1-4 (eGFR 15-90 mL/min/1.73 m²) for at least 3 months.
  * Willing and able to provide informed consent

Exclusion Criteria:

* • Patients with end-stage renal disease (CKD stage 5 or on dialysis).

  * History of kidney transplantation.
  * Acute kidney injury within the past 3 months.
  * Pregnant or lactating women.
  * Patients with severe comorbid conditions (e.g., active malignancy, severe heart failure).
  * Use of medications known to significantly affect renal function (other than standard antihypertensive or antidiabetic therapy).

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults aged above 18 years with chronic kidney disease stages 1-4 and type 2 Diabetes Milletus
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the influence of dietary pattern on the progression of chronic kidney disease among patients with type 2 Diabetes Milletus | 6 month
  Primary Outcomes Measures
  1. change in estimated glomerular filtration rate (eGFR) from baseline to 6 month using CKD-EPI formula mL/min/1.73 m² Time frame 6 month